CLINICAL TRIAL: NCT02824861
Title: Bemobile: A Text Intervention to Support Physical Activity in Cancer Survivors
Brief Title: Bemobile Intervention to Support Physical Activity in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Nancy Gell, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHRMS15-405; VCC1504 (Other: Vermont Cancer Center)
Record Dates: First submitted 2016-07-02; First posted 2016-07-07 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Intervention (Experimental): Participants receive text messages to a personal cell phone over 8 weeks, wear a fitbit to monitor physical activity, and communicate with a health coach intermittently over 2 weeks
  Interventions: Behavioral: Bemobile
- Active Control (Active Comparator): Participants receive and wear a fitbit only for 8 weeks
  Interventions: Behavioral: Bemobile

INTERVENTIONS:
Behavioral: Bemobile

SUMMARY:
This study evaluates a technology based intervention (physical activity tracker, text messages, health coach, global positioning system enabled location based feedback on physical activity) to support physical activity in cancer survivors after completing oncology rehabilitation. In Phase 1 all participants received the full intervention. In phase II participants are randomly assigned to receive the full intervention or a fitbit only.

DETAILED DESCRIPTION:
This intervention, offered to participants after completing oncology rehabilitation, integrates known preferences and determinants of physical activity participation in women and breast cancers survivors including social support, professional guidance, self-efficacy, goal setting, self-regulation, and environmental awareness delivered through accessible technology. For the iteration phase, the investigators will conduct an initial, abbreviated intervention wave lasting 4 weeks; the investigators will then incorporate participant input and feedback on the specific components to refine the intervention prior to a pilot trial. Means of delivering the components include communication and support through tailored text messaging, health coaching phone calls, self-monitoring of physical activity through a wearable sensor, and environmental assessment of community physical activity options (e.g., parks, fitness centers, trails) based on global positioning system information.

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis
* Impending graduation from oncology rehabilitation

Exclusion Criteria:

* Metastatic cancer
* Concurrent radiation or chemotherapy
* No cell phone
* Inability to read or speak English.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Step counts | 8 weeks
  Mean daily step counts as assessed by Actigraph Accelerometer
Change from Baseline in Moderate to Vigorous Physical Activity (MVPA) | 8 weeks
  Weekly accumulated minutes spent in MVPA as assessed by Actigraph Accelerometer

SECONDARY OUTCOMES:
Change in Weekly average of mean daily step counts | 8 weeks
  Step counts assessed during the intervention with the Fitbit One
Change from Baseline in Self-efficacy to perform exercise | 8 weeks
  Scale developed by Garcia and King
Change from Baseline in Self-regulation | 8 weeks
  Scale Developed R. Umstattd
Change from Baseline in Fatigue | 8 weeks
  Fatigue Symptom Inventory (FSI)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available